CLINICAL TRIAL: NCT02320110
Title: Correlation of Circulating Irisin and Adipokine Levels Across a Broad Spectrum of Body Mass Index Ranging From Undernourished to Obese and With Insulin Resistance and Risk Factors for the Metabolic Syndrome in Hispanic Children
Brief Title: Correlation of Irisin and Adipokine Levels With Body Mass Index and Risk Factors for Metabolic Syndrome in Hispanic Children
Status: Completed | Type: Observational
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Leticia Elizondo-Montemayor, Dean of the Clinical Nutrition and Obesity Research Center. School of Medicine TEC Salud. Tecnológico de Monterrey., Instituto Tecnologico y de Estudios Superiores de Monterey
Other Study IDs: DIETARYHABITS2014-CINCO
Record Dates: First submitted 2014-12-02; First posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Obesity; Thinness
Keywords: Irisin; Adiponectin; Leptin; Insulin resistance; Body Mass Index; Obesity; Metabolic Syndrome; Lipid Profile; Diabetes Mellitus
MeSH Terms: conditions — Overweight; Obesity; Thinness; Insulin Resistance; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Childhood obesity is one of the most serious global public health challenges of the 21st century (Daniels et al., 2009). Mexico has the highest prevalence of obesity, (Secretaría de Salud, 2009); 34.4% of children and 35% of adolescents are overweight or obese (ENSANUT 2012). Obesity has major health consequences for children and adolescents; On the other hand, undernutrition as well has important deleterious consequences on children's health.

Anything that disrupts energy balance may cause individuals to be underweight, overweight or obese. Fat has been considered an endocrine organ for some time (Elizondo, 2011). Recently, skeletal muscle has been shown to function as a peripheral endocrine organ by releasing myokines, (Pedersen, 2012). Most recently, a new identified hormone secreted by muscle tissue in mouse, irisin, has been discovered. Irisin acts on white adipose cells in culture and in vivo to stimulate UCP1 expression and a broad program of brown-fat-like development. Irisin was induced with exercise in mice and humans which caused an increase in energy expenditure in mice with no changes in movement or food intake (Boström et al., 2012).

Irisin was thus, promptly hypothesized as a hormone influencing body weight, obesity and type 2 diabetes mellitus, among other conditions (Sanchis-Gomar et al., 2012). Some studies have indicated that circulating levels of irisin in humans correlate positively with anthropometric parameters such as BMI, fat mass, fat free mass, and are higher in obese patients compared to lean ones (Stengel et al., 2013; Huh et al., 2012; Roca-Rivada et al., 2013; Crujeiras et al., 2014; Pardo, 2014). Studies have shown an association between irisin levels, insulin resistance and the metabolic syndrome (Park et al., 2013; de la Iglesia et al., 2014; Crujeiras et al., 2014; Pardo et al., 2014). However, some others have found a negative correlation with anthropometric parameters, finding lower irisin levels in obese patients (Moreno-Navarrete et al., 2013). Noteworthy, all these studies have been performed in adults. To date, there are only two studies evaluating irisin levels in children. One found that a 1-year long lifestyle intervention program was associated with an elevation in irisin levels in obese children, although no correlation was found between irisin levels and anthropometric markers (Blüher et al., 2014). The other study investigated normal weight Saudi children and found correlations between circulating irisin and glucose and HDLc, but a negative association with insulin resistance (Al-Daghri et al, 2014).

Besides, associations between irisin levels and adiponectin, leptin and resistin in the set of obesity have been explored, the three of them are implicated in the physiopatology of obesity.

As there are still conflicting data regarding the association of irisin with anthropometric parameters, obesity and the metabolic syndrome, as well as its 'association with other adiponectines, and most important, there is scarce data of these associations in children, the objective of this study will be to correlate the circulating irisin and adipokines levels across a broad spectrum of body mass index ranging from undernourished to obese as well as with insulin resistance and risk factors for the metabolic syndrome in Hispanic children.

The sample size with statistical power for this study yielded a sample of 40 children. Frozen stored plasma (-80°C) will be taken from a previous study performed in children which has been published (Elizondo-Montemayor et al., 2014). The samples will be divided into five groups, 8 per group, according to the CDC and American Academy of Pediatrics body mass index percentile classification: 1.) underweight = <3 percentile; 2.) normal weight = >3 - < 85 percentile; 3.) Overweight = >85 - < 95 percentile, and 4.) obese = > 95 percentile. The fifth group will correspond to children with known metabolic syndrome according to the classification specified by Cooks et al (2008). Anthropometric measurements will include BMI, percentile BMI, waist circumference, % body fat, fat mass, fat free mass, and triceps skin fold. Biochemical measurements will include glucose, total cholesterol, low-density cholesterol (LDL), high-density cholesterol (HDL-c) and triglycerides. Clinical measurements will include blood pressure, physical activity records and dietary habits. All biochemical, anthropometric and clinical measurements were previously performed in a former published study (Elizondo-Montemayor et al., 2014).

Irisin, adiponectin and leptin will be measured in plasma media using commercial ELISA kits.

DETAILED DESCRIPTION:
Background Childhood obesity is one of the most serious global public health challenges of the 21st century (Daniels et al., 2009). Mexico has the highest prevalence of obesity, worldwide; 34.4% of children and 35% of adolescents are overweight or obese (ENSANUT 2012). Among other complications, overweight and obese children are predisposed to develop dyslipidemias, hypertension, the metabolic syndrome (MetS) and non-alcoholic fatty liver disease at a younger age, as well as to become obese as adults (Daniels et al., 2009; Elizondo-Montemayor et al., 2010). On the other hand, undernutrition in children conveys to very detrimental health effects such as stunting, puberty retardation, motor retardation (Roulet et al., 2005), osteoporosis and fractures (Saunders et al., 2011), immunologic deficit, and altered function of every organ and system, such as the heart, lungs, kidneys, gastrointestinal tract and the nervous system, among others (Lecours et al, 2001; Saunders et al., 2011).

A balance between energy intake and energy expenditure is required to sustain a normal body weight. Anything that disrupts this balance may cause individuals to be underweight, overweight or obese. Diverse signals, central and peripheric participate in the regulation of energy balance. Fat has been considered an endocrine organ due to the many peptides and hormones that it secrets that act upon peripheral and central tissues, and their contribution to insulin resistance or sensitivity and body weight regulation among other functions (Elizondo, 2011). Recently, skeletal muscle has been shown to function as a peripheral endocrine organ by releasing myokines, peptide signals, which are implicated in the regulation of metabolic pathways (Pedersen and Febbraio, 2012). Most recently, a new identified hormone secreted by muscle tissue in mouse, irisin, has been discovered. Irisin acts on white adipose cells in culture and in vivo to stimulate UCP1 expression and a broad program of brown-fat-like development. In mouse, PGC1alfa expression in muscle stimulates increase in expression of FNDC5, a membrane protein that is cleaved and secreted as this novel hormone, irisin. Irisin is induced with exercise in mice and humans, and medley increased irisin levels in blood cause an increase in energy expenditure in mice with no changes in movement or food intake (Boström et al., 2012).

Irisin was thus, promptly hypothesized as a hormone influencing body weight, obesity and type 2 diabetes mellitus, among other conditions (Sanchis-Gomar et al., 2012). Some studies have indicated that circulating levels of irisin in humans correlate positively with anthropometric parameters such as BMI, fat mass, fat free mass, and are higher as these parameters increase, this is, irisin levels are higher in obese patients compared to lean ones (Stengel et al., 2013; Huh et al., 2012; Roca-Rivada et al., 2013; Crujeiras et al., 2014; Pardo et al., 2014). Studies have shown an association between irisin levels, insulin resistance and the metabolic syndrome (Park et al., 2013; de la Iglesia et al., 2014; Crujeiras et al., 2014; Pardo et al., 2014). However, some others have found a negative correlation with anthropometric parameters, finding lower irisin levels in obese patients (Moreno-Navarrete et al., 2013). Noteworthy, all these studies have been performed in adults in different circumstances or diseased states. To date, there are only two studies evaluating irisin levels in children. One found that a 1-year long lifestyle intervention program was associated with improvement in anthropometric and metabolic parameters and led to an elevation in irisin levels in obese children, although no correlation was found between irisin levels and anthropometric markers (Blüher et al., 2014). The other study investigated normal weight Saudi children and found correlations between circulating irisin and glucose and HDLc, but a negative association with insulin resistance (Al-Daghri et al., 2014).

Besides, associations between irisin levels and adiponectin, leptin and resistin in the set of obesity have been explored. Leptin plays a pivotal role in regulating energy homeostasis, food intake and many neuroendocrine functions, specially triggering puberty in children. Leptin is increased in obese patients, associated with a leptin-resistant state (Blüher and Mantzoros, 2009). Adiponectin is an insulin sensitizing hormone; obese patients have lower levels than normal-weight ones. Circulating adiponectin levels are low in central obesity (Dalamaga et al., 2012), and this low level has been associated with the metabolic syndrome across all ages (Siitonen et al., 2011). Resistin has been associated with insulin resistance, and recently as a proinflamatory adipocytokine (McTernan et al., 2006). Some studies have found a negative correlation between irisin and adiponectin levels (Park et al., 2013), while other have found no association either with leptin or adiponectin (Blüher et al., 2014) here are still conflicting data regarding the association of irisin with anthropometric parameters, obesity and the metabolic syndrome, as well as its 'association with other adipokines, and most important, there is scarce data of these associations in children, the objective of this study will be to correlate the circulating irisin and adipokines levels across a broad spectrum of body mass index ranging from undernourished to obese as well as with insulin resistance and risk factors for the metabolic syndrome in Hispanic children.

There is still conflicting data regarding the association of irisin with anthropometric parameters, obesity and the metabolic syndrome, as well as its 'association with other adipokines, and most important, there is scarce data of these associations in children. Therefore, the objective of this study will be to correlate the circulating irisin and adipokines levels across a broad spectrum of body mass index ranging from undernourished to obese as well as with insulin resistance and risk factors for the metabolic syndrome in Hispanic children.

Study Population The population was previously described. (Elizondo-Montemayor et al., 2014) An open invitation was made to school-aged children from eight public schools representative of all geographical areas of Monterrey, the second largest city in México. Children that accepted the invitation were randomly selected and screened according to BMI percentiles. The sample size is 40 children. The population will be divided into five groups, 8 per group. Four of the groups will be divided according to the CDC body mass index percentiles: 1.) underweight = <3percentile; 2.) normal weight = >3 - < 85 percentile; 3.) Overweight = >85 - < 95 percentile, and 4.) obese = > 95 percentile. The fifth group will correspond to children with known metabolic syndrome.

Signed consent was obtained from both parents/care givers and children. Approvals by the Ethics and Research Committees of the School of Medicine Tecnológico de Monterrey and by the State Health Secretariat, as well as by the Education Authorities were obtained. Participants did not receive gratification during the study.

Anthropometric and Clinical Evaluation Anthropometric measurements were performed in all participants at each school. Height was determined to the nearest 0.5 cm (portable Seca® stadiometer, North America) and weight to the nearest 0.1 kg while children wore light clothing, no socks or shoes (TANITA TBF 300® scale, Arlington, Illinois). Percentage of body fat (%BF) was measured by bioimpedance (same TANITA scale). WC was measured to the nearest 0.1 cm at the level of the umbilicus with a flexible fiberglass tape while the subjects were standing, after gently exhaling, and with no clothing on the area. Tricipital skin fold (TSF) was measured using a Lange skinfold caliper. BMI was calculated by weight-kilograms divided by the square of height-meters. Fat mass and fat free mass were calculated according to the specific predetermined formulas. Measurements were performed at the same time each day by the same three trained registered dietitians (RD) in all children to control the inter-observer variability. Blood pressure was measured by the same physician, using an aneroid sphygmomanometer (Welch-Allyn®) following the American Heart Association (AHA) technique; two measurements were obtained while participants were calmed and seated.

Laboratory Assessment Blood samples were taken after a 12-hour overnight fast and were kept at 2 to 8°C and centrifuged within the first 3 hours. Serum total cholesterol (TC), HDL-C, low-density lipoprotein cholesterol (LDL-C), triglycerides (TG), and glucose were measured by reflective photometry (Beer-Lambert's law) using an automated analyzer (Architect c8000; Abbott Laboratories, Abbott Park, IL), with an intra- and inter-assay coefficient variation below 4.7%. Plasma samples were then stored at -80°C. Irisin, adiponectin, insulin and leptin will be measured in plasma media using commercial ELISA kits. The assays will be conducted in 96-well microplates according to the manufacturer's instructions (Irisin, adiponectin, insulin and leptin ELISA kit; Phoenix Pharmaceuticals, Inc., Burlingame, CA, USA). Absorbance from each sample will measured in duplicate using a spectrophotometric microplate reader at wavelength of 450 nm (BioTek Instruments, Winooski, VT, USA).

Statistical Methods MINITAB version 16 (Minitab Inc., State College, PA, USA) will be used to analyze the differences between anthropometric and biochemical parameters and irisin levels; Microsoft Excel 2007 (Microsoft Corp., Redmond, WA, USA) will be used to incorporate the input of data. The results will be expressed as mean ± standard deviation (s.d.), as absolute number or as percentage (%) and their corresponding 95% confidence intervals (CI). Comparisons between groups for the dependent variables will be made using paired Student´s t-test for means and McNemar test for proportions. For independent variables, the normality will be revised both, graphically and by the Shapiro-Wilk test, and subsequently, the comparisons between groups will be determined using z-test. To assess the association between anthropometric, clinical and biochemical variables and irisin levels, a simple linear regression will be used. The mean comparisons between gender groups will be determined using t-test for independent samples. All tests will be interpreted based on two-tailed hypothesis. The significance level will be set at 0.05 in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Attendance to school from first to sixth grade
* Ages 6-12 years
* Hispanic origin
* Both parents Hispanic
* 12 hour overnight fast
* Signed consent from both parents/care givers and active assent from children

Exclusion Criteria:

* Disapproval by the children's physician due to any at-risk medical condition known by the parents
* Use of drugs for high blood pressure, hyperglycemia, or dyslipidemia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Obese, overweight, normal weight and underweight Hispanic, school-aged children from eight public schools representative of Monterrey, the second largest city in México.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Irisin levels identification in Hispanic children | 3 months
Correlation of irisin levels with body mass index percentiles in Hispanic children | 3 months
  Correlation of irisin plasma levels with body mass index percentiles
Correlation of irisin leves with risk factors for metabolic syndrome in Hispanic children | 3 months
  The risk factors include: waist circumference, % body fat, triceps skin fold, fat mass, fat free mass and blood presurre measurements, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides and glucose serum levels

SECONDARY OUTCOMES:
Irisin plasma levels and adiponectin, leptin, insulin and resistin. | 3 months
  correlation of irisin plasma levels adiponectin, leptin, resistin and insluin

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Elizondo-Montemayor, MD, Principal Investigator — Clinical Nutrition and Obesity Research Center. TEC Salud, School of Medicine Tecnológico de Monterrey
Locations (1):
- Clinical Nutrition and Obesity Research Center. School of Medicine, TEC Salud, Tecnológico de Monterrey, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Daniels SR, Jacobson MS, McCrindle BW, Eckel RH, Sanner BM. American Heart Association Childhood Obesity Research Summit Report. Circulation. 2009 Apr 21;119(15):e489-517. doi: 10.1161/CIRCULATIONAHA.109.192216. Epub 2009 Mar 30. No abstract available. PMID 19332458
- [Background] Elizondo-Montemayor L, Serrano-Gonzalez M, Ugalde-Casas PA, Cuello-Garcia C, Borbolla-Escoboza JR. Metabolic syndrome risk factors among a sample of overweight and obese Mexican children. J Clin Hypertens (Greenwich). 2010 May;12(5):380-7. doi: 10.1111/j.1751-7176.2010.00263.x. PMID 20546382
- [Background] Roulet M, Cheseaux M, Coti P. Consequences of disease-related malnutrition in children and adolescents: Mortality, morbidity and costs. Arch Pediatr 12(4): 207-213, 2005
- [Background] Secretaría de Salud. México avanza en la cobertura universal de salud: Felipe Calderón. México Sano. 2009;8:3.
- [Background] Saunders J, Smith T, Stroud M. Malnutrition and undernutrition. Medicine 39(1): 45-50, 2011
- [Background] Lecours AR, Mandujano M, Romero G. Ontogeny of brain and cognition: relevance to nutrition research. Nutr Rev. 2001 Aug;59(8 Pt 2):S7-11; discussion S11-2. doi: 10.1111/j.1753-4887.2001.tb05504.x. No abstract available. PMID 11519671
- [Background] Elizondo, L. Hernández, C. Zamora, M. (2011). Terapia Nutricia Médica en Ginecología y Obstetricia. México: McGraw-Hill.
- [Background] Pedersen BK, Febbraio MA. Muscles, exercise and obesity: skeletal muscle as a secretory organ. Nat Rev Endocrinol. 2012 Apr 3;8(8):457-65. doi: 10.1038/nrendo.2012.49. PMID 22473333
- [Background] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023
- [Background] Sanchis-Gomar F, Lippi G, Mayero S, Perez-Quilis C, Garcia-Gimenez JL. Irisin: a new potential hormonal target for the treatment of obesity and type 2 diabetes. J Diabetes. 2012 Sep;4(3):196. doi: 10.1111/j.1753-0407.2012.00194.x. No abstract available. PMID 22372821
- [Background] Stengel A, Hofmann T, Goebel-Stengel M, Elbelt U, Kobelt P, Klapp BF. Circulating levels of irisin in patients with anorexia nervosa and different stages of obesity--correlation with body mass index. Peptides. 2013 Jan;39:125-30. doi: 10.1016/j.peptides.2012.11.014. Epub 2012 Dec 3. PMID 23219488
- [Background] Huh JY, Panagiotou G, Mougios V, Brinkoetter M, Vamvini MT, Schneider BE, Mantzoros CS. FNDC5 and irisin in humans: I. Predictors of circulating concentrations in serum and plasma and II. mRNA expression and circulating concentrations in response to weight loss and exercise. Metabolism. 2012 Dec;61(12):1725-38. doi: 10.1016/j.metabol.2012.09.002. Epub 2012 Sep 25. PMID 23018146
- [Background] Roca-Rivada A, Castelao C, Senin LL, Landrove MO, Baltar J, Belen Crujeiras A, Seoane LM, Casanueva FF, Pardo M. FNDC5/irisin is not only a myokine but also an adipokine. PLoS One. 2013 Apr 11;8(4):e60563. doi: 10.1371/journal.pone.0060563. Print 2013. PMID 23593248
- [Background] Crujeiras AB, Zulet MA, Lopez-Legarrea P, de la Iglesia R, Pardo M, Carreira MC, Martinez JA, Casanueva FF. Association between circulating irisin levels and the promotion of insulin resistance during the weight maintenance period after a dietary weight-lowering program in obese patients. Metabolism. 2014 Apr;63(4):520-31. doi: 10.1016/j.metabol.2013.12.007. Epub 2013 Dec 18. PMID 24439241
- [Background] Pardo M, Crujeiras AB, Amil M, Aguera Z, Jimenez-Murcia S, Banos R, Botella C, de la Torre R, Estivill X, Fagundo AB, Fernandez-Real JM, Fernandez-Garcia JC, Fruhbeck G, Gomez-Ambrosi J, Rodriguez R, Tinahones FJ, Fernandez-Aranda F, Casanueva FF. Association of irisin with fat mass, resting energy expenditure, and daily activity in conditions of extreme body mass index. Int J Endocrinol. 2014;2014:857270. doi: 10.1155/2014/857270. Epub 2014 Apr 22. PMID 24864142
- [Background] Park KH, Zaichenko L, Brinkoetter M, Thakkar B, Sahin-Efe A, Joung KE, Tsoukas MA, Geladari EV, Huh JY, Dincer F, Davis CR, Crowell JA, Mantzoros CS. Circulating irisin in relation to insulin resistance and the metabolic syndrome. J Clin Endocrinol Metab. 2013 Dec;98(12):4899-907. doi: 10.1210/jc.2013-2373. Epub 2013 Sep 20. PMID 24057291
- [Background] de la Iglesia R, Lopez-Legarrea P, Crujeiras AB, Pardo M, Casanueva FF, Zulet MA, Martinez JA. Plasma irisin depletion under energy restriction is associated with improvements in lipid profile in metabolic syndrome patients. Clin Endocrinol (Oxf). 2014 Aug;81(2):306-11. doi: 10.1111/cen.12383. Epub 2014 Jan 7. PMID 24325584
- [Background] Moreno-Navarrete JM, Ortega F, Serrano M, Guerra E, Pardo G, Tinahones F, Ricart W, Fernandez-Real JM. Irisin is expressed and produced by human muscle and adipose tissue in association with obesity and insulin resistance. J Clin Endocrinol Metab. 2013 Apr;98(4):E769-78. doi: 10.1210/jc.2012-2749. Epub 2013 Feb 22. PMID 23436919
- [Background] Bluher S, Panagiotou G, Petroff D, Markert J, Wagner A, Klemm T, Filippaios A, Keller A, Mantzoros CS. Effects of a 1-year exercise and lifestyle intervention on irisin, adipokines, and inflammatory markers in obese children. Obesity (Silver Spring). 2014 Jul;22(7):1701-8. doi: 10.1002/oby.20739. Epub 2014 Mar 25. PMID 24644099
- [Background] Al-Daghri NM, Alkharfy KM, Rahman S, Amer OE, Vinodson B, Sabico S, Piya MK, Harte AL, McTernan PG, Alokail MS, Chrousos GP. Irisin as a predictor of glucose metabolism in children: sexually dimorphic effects. Eur J Clin Invest. 2014 Feb;44(2):119-24. doi: 10.1111/eci.12196. Epub 2013 Dec 6. PMID 24188288
- [Background] Bluher S, Mantzoros CS. Leptin in humans: lessons from translational research. Am J Clin Nutr. 2009 Mar;89(3):991S-997S. doi: 10.3945/ajcn.2008.26788E. Epub 2009 Jan 28. PMID 19176740
- [Background] Dalamaga M, Diakopoulos KN, Mantzoros CS. The role of adiponectin in cancer: a review of current evidence. Endocr Rev. 2012 Aug;33(4):547-94. doi: 10.1210/er.2011-1015. Epub 2012 Apr 30. PMID 22547160
- [Background] Siitonen N, Pulkkinen L, Lindstrom J, Kolehmainen M, Eriksson JG, Venojarvi M, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Tuomilehto J, Uusitupa M. Association of ADIPOQ gene variants with body weight, type 2 diabetes and serum adiponectin concentrations: the Finnish Diabetes Prevention Study. BMC Med Genet. 2011 Jan 10;12:5. doi: 10.1186/1471-2350-12-5. PMID 21219602
- [Background] McTernan PG, Kusminski CM, Kumar S. Resistin. Curr Opin Lipidol. 2006 Apr;17(2):170-5. doi: 10.1097/01.mol.0000217899.59820.9a. PMID 16531754